CLINICAL TRIAL: NCT01192126
Title: A Study to Evaluate the Product Performance of a Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 662
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-11

CONDITIONS: Myopia; Contact Lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch & Lomb new daily disposable (Experimental): New daily disposable contact lenses
  Interventions: Device: Bausch & Lomb new daily disposable
- Johnson & Johnson Acuvue Moist (Active Comparator): Contact lenses
  Interventions: Device: Johnson & Johnson Acuvue Moist

INTERVENTIONS:
Device: Bausch & Lomb new daily disposable — Test lenses are to be worn for approximately one week. Lenses will be worn on a daily wear basis.
  Arms: Bausch & Lomb new daily disposable
Device: Johnson & Johnson Acuvue Moist — Control lenses are to be worn for approximately one week. Lenses will be worn on a daily wear basis.
  Arms: Johnson & Johnson Acuvue Moist

SUMMARY:
The objective of the study is to evaluate the product performance of visual acuity of the Bausch + Lomb investigational daily disposable contact lenses compared to the currently marketed Johnson & Johnson Acuvue Moist contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adapted soft contact lens wearers that are interested in daily disposable wear or currently adapted daily disposable soft contact lens wearers.
* Subjects must agree to wear study lenses on a daily disposable basis for approximately one week and crossover to wear another study lens for one week.
* Subjects must be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
* Subjects must have clear central corneas that are free of any anterior segment disorders.
* Subjects must be myopic and require lens correction from -1.00 D to -6.00 diopters (D) in each eye.

Exclusion Criteria:

* Subjects who have worn gas permeable contact lenses within the last 30 days or who have worn polymethylmethacrylate lenses within the last 3 months.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an affect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects who are not correctable to 32 letters (0.3 logMAR) in each eye with soft spherical contact lenses.
* Subjects who currently wear monovision, multifocal, or toric contact lenses.
* Subjects with an ocular astigmatism of 1.00 D or greater in either eye.
* Subjects with anisometropia (spherical equivalent) of greater than 1.00 D.
* Subjects with any grade 2 or greater finding during the slit lamp examination (refer to Appendix B for methods of clinical evaluation).
* Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Subjects with any "Present" finding during the slit lamp examination (refer to Appendix B for methods of clinical evaluation) that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study.
* Subjects who are aphakic.
* Subjects who are amblyopic.
* Subjects who have presbyopia.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who are allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bev Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two week, multicenter, open label, bilateral, crossover study. First Participant was enrolled 08/23/2010 and last participant exited the study 10/08/2010.
Pre-assignment Details: 102 participants(204 eyes) were enrolled in this study.
Groups:
- B & L Daily Disposable Lens, Then J & J Acuvue Moist: Bausch & Lomb new daily disposable lenses are to be worn for approximately one week. Crossover to Johnson & Johnson Acuvue Moist lenses to be worn for approximately one week. Lenses will be worn on a daily wear basis.
- J & J Acuvue Moist, Then B & L Daily Disposable Lens: Johnson & Johnson Acuvue Moist lenses are to be worn for approximately one week. Crossover to Bausch & Lomb new daily disposable lenses to be worn for approximately one week. Lenses will be worn on a daily wear basis.
Period: First Intervention (1 Week)
Arm/Group | B & L Daily Disposable Lens, Then J & J Acuvue Moist | J & J Acuvue Moist, Then B & L Daily Disposable Lens
Started | 51 | 51
Completed | 49 | 50
Not Completed | 2 | 1
Not completed — Unacceptable Distance Visual Acuity | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Period: Second Intervention (1 Week)
Arm/Group | B & L Daily Disposable Lens, Then J & J Acuvue Moist | J & J Acuvue Moist, Then B & L Daily Disposable Lens
Started | 49 | 50
Completed | 49 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Overall Study: All eligible subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Distance High contrast logMAR visual acuity (VA), difference between the test and control lens at dispensing visit and 1 week follow-up, crossover visit and 1 week follow-up.
Time Frame: Dispensing Visit and 1 week follow-up
Population: All Eligible Dispensed Eyes
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Bausch & Lomb New Daily Disposable: New daily disposable contact lenses
  Bausch & Lomb new daily disposable : Test lenses are to be worn for approximately one week. Lenses will be worn on a daily wear basis.
- Johnson & Johnson Acuvue Moist: Contact lenses
  Johnson & Johnson Acuvue Moist : Control lenses are to be worn for approximately one week. Lenses will be worn on a daily wear basis.
Arm/Group | Bausch & Lomb New Daily Disposable | Johnson & Johnson Acuvue Moist
Number analyzed (Participants) | 99 | 99
Number analyzed (eyes) | 198 | 198
LogMAR
  Dispensing Visit | -0.056 (0.079) | -0.070 (0.066)
  1 Week Follow-up | -0.063 (0.079) | -0.065 (0.079)

2. Primary Outcome: Slit Lamp Examination > Grade 2
Description: Slit lamp findings for each eye will be assessed at each study visit, including epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates, will be graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). Slit lamp > 2.
Time Frame: All study visits from screening through 2 week follow-up
Population: All Dispensed Eyes
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb New Daily Disposable | Johnson & Johnson Acuvue Moist
Number analyzed (Participants) | 99 | 99
Number analyzed (eyes) | 198 | 198
Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Bausch & Lomb New Daily Disposable | Johnson & Johnson Acuvue Moist
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other